CLINICAL TRIAL: NCT00395850
Title: Disulfiram for Cocaine Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-13441; 5R01DA013441-02 (NIH); 5R01DA013441-03 (NIH); 5R01DA013441-04 (NIH); 5R01DA013441-06 (NIH); 1R01DA013441-01A1 (NIH); 7R01DA013441-05 (NIH); 5R01DA013441-09 (NIH); 5R01DA013441-10 (NIH); 5R01DA013441-08 (NIH); R01DA013441 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-09

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; disulfiram; clinical trial; methadone maintenance; pharmacogenetics; dopamine beta-hydroxylase
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Disulfiram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): microcrystalline cellulose
  Interventions: Drug: Disulfiram
- 2 (Experimental): disulfiram at 250 mg/day
  Interventions: Drug: Disulfiram
- 3 (Experimental): Disulfiram at 375 mg/day
  Interventions: Drug: Disulfiram
- 4 (Experimental): Disulfiram at 500 mg/day
  Interventions: Drug: Disulfiram

INTERVENTIONS:
Drug: Disulfiram — Disulfiram at 0, 250, 375, or 500 mg/day for 12 weeks

SUMMARY:
This study examines the influence of dopamine beta-hydroxylase enzyme activity on the clinical efficacy of the novel pharmacotherapy, disulfiram, for treating cocaine dependence in cocaine-dependent patients, some of whom are opioid dependent and maintained on an FDA-approved opioid agonist. Cocaine dependence as well as co-morbid cocaine and opioid-dependence is associated with more public health issues and poorer treatment prognosis when admitted to methadone maintenance. Yet no effective pharmacotherapies have been developed to treat cocaine dependence to date. One novel pharmacotherapy, disulfiram, has shown some promise as a treatment for this disorder in several clinical trials at a dose of 250 mg/day or more (e.g., Carroll et al., 1998, 2004). This 14-week, randomized, double blind clinical trial will provide treatment for up to160 cocaine-dependent individuals, aged 18-65 years. Participants who are opioid dependent will be stabilized on methadone maintenance during the first 2 weeks and baseline cocaine use will be assessed; participants will be stratified by DBH genotype and randomly assigned to receive disulfiram at either 0, 250, 375 or 500 mg/day. During induction onto methadone for opioid dependent individuals, participants are administered increasing doses of methadone on a daily basis until maintenance doses are attained. At the beginning of week 3, participants receive methadone, if relevant, plus disulfiram or placebo disulfiram according to their randomized assignments, and are maintained on study medication(s) through week 14. At the end of the study, participants will undergo detoxification from the opioid agonist, if relevant, and active/placebo medication over a 4- to 6-week period. All participants receive weekly 1-hour psychotherapy (Cognitive Behavioral Treatment) with experienced clinicians specifically trained to deliver the therapy and who will receive ongoing supervision. Participants undergo a delay discounting session during week 1. The primary outcomes will be retention, reduction in opioid and cocaine use, as assessed by self-report and confirmed by thrice-weekly urinalyses, and disulfiram side-effects profile. Secondary outcomes will include reductions in other illicit drug and alcohol use, and improvements in psychosocial functioning. The prognostic relevance of genotype at the DBH locus, DβH activity, etc., on response to disulfiram will be examined.

ELIGIBILITY:
Inclusion Criteria:

* current users of cocaine, including having a cocaine-positive urine
* self-reported use of > 7 gm during the preceding 6 months and > 1 time/week in at least one month preceding study entry
* meet DSM-IV criteria for cocaine dependence

Exclusion Criteria:

* current diagnosis of alcohol dependence
* significant medical conditions such as abnormal liver function
* active hepatitis
* hypertension
* a current cardiac condition or high risk of cardiovascular disease
* seizure disorders
* any another significant underlying medical condition which would contraindicate disulfiram or methadone treatment
* meeting DSM-IV psychiatric classifications for schizophrenia, bipolar disorder, or other psychotic disorders
* exhibiting current suicidality or homicidality
* pregnancy
* current use of a prescribed psychotropic medication (e.g., antidepressants, anxiolytics, antipsychotics, anticonvulsants, etc.) which cannot be discontinued current use of medications such as anticoagulants, isoniazid, metronidazole, clotrimazole, and paraldehyde.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2007-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 2006 and September 2011. Opioid- or nonopioid dependent treatment seekers recruited via newspaper ads, radio ads, flyer, word-of-mouth and referrals and attended the Treatment Research Unit, initially located in an off-campus facility and then relocated to the the Psychiatric Research Institute (12/08).
Pre-assignment Details: Participants underwent either a two-week induction onto methadone (if opioid dependent) or a two-week baseline period prior to randomization to the treatment arms and receiving medication starting in week 3. Those receiving at >1 dose of medication and completing assessments at at least 2 time points during week 3 were include in the analyses.
Groups:
- Placebo: microcrystalline cellulose
- Disulfiram 250: disulfiram at 250 mg/day
- Disulfiram 375: Disulfiram at 375 mg/day
- Disulfiram 500: Disulfiram at 500 mg/day
Period: Pre-randomization Baseline/Induction
Arm/Group | Placebo | Disulfiram 250 | Disulfiram 375 | Disulfiram 500
Started | 118 (Pre-randomization and disulfiram (disulf) administration) | 0 | 0 | 0
Completed | 107 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0
Not completed — noncompliance (missed med/urine) | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Not completed — Inconsistent attendance | 1 | 0 | 0 | 0
Period: Randomization to Disulfiram/ Pre-admin
Arm/Group | Placebo | Disulfiram 250 | Disulfiram 375 | Disulfiram 500
Started | 27 | 25 | 30 | 25
Completed | 22 | 23 | 24 | 21
Not Completed | 5 | 2 | 6 | 4
Not completed — noncompliance - missed med/urines | 2 | 2 | 6 | 4
Not completed — noncompliance with alcohol use | 1 | 0 | 0 | 0
Not completed — suicidal ideation | 1 | 0 | 0 | 0
Not completed — work schedule conflict | 1 | 0 | 0 | 0
Period: Disulfiram/Placebo Treatment
Arm/Group | Placebo | Disulfiram 250 | Disulfiram 375 | Disulfiram 500
Started | 20 (Received >= 1 disulfiram dose. Two baseline/randomized subjects dropped out before receiving disulf) | 23 (Received at least one dose of disulfiram) | 24 (Received at least one dose of disulfiram) | 21 (Received at least one dose of disulfiram)
Completed | 11 | 9 | 5 | 8
Not Completed | 9 | 14 | 19 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Disulfiram 250 | Disulfiram 375 | Disulfiram 500 | Total
Number analyzed (Participants) | 27 | 25 | 30 | 25 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 25 | 30 | 25 | 107
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.0 (12.4) | 39.8 (11.3) | 39.4 (10.1) | 40.4 (10.1) | 40.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 13 | 8 | 41
  Male | 17 | 15 | 17 | 17 | 66
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 30 | 25 | 107

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use Over Time
Description: Urine toxicology results (dichotomous: positive or negative) for the presence of cocaine/cocaine metabolite during the disulfiram phase of the study. The change in the probability of a cocaine positive urine sample per day was assessed for each dose compared with placebo and slopes for each dose condition were calculated from Repeated Measures Genearlized Linear Models on a Binomial distribution (thus a Repeated Measures Logistic Regression)
Time Frame: thrice weekly for 12 weeks
Population: number is based on those who participated long enough to have assessments completed at two time points during the disulfiram phase
Measure: Number; unit: slope (change in prob of coc-pos utox/d)
Arm/Group | Placebo | Disulfiram 250 | Disulfiram 375 | Disulfiram 500
Number analyzed (Participants) | 27 | 25 | 30 | 25
slope (change in prob of coc-pos utox/d) | 0.01 | 0.007 | -0.01 | 0.007
Statistical Analysis 1: Comparison: Disulfiram 250 vs Disulfiram 375 vs Disulfiram 500; Used placebo group as contrast to determine whether slopes of disulfiram groups differed from slope of placebo group data; Test type: Superiority or Other; p < 0.05, Repeated Measures Logistic Regression; Repeated Measures Generalized Linear Models on a Binomial distribution, thus a Repeated Measures Logistic Regression; Slope = -1.02

2. Secondary Outcome: Retention
Time Frame: 14 weeks
Population: those who were entered the disulfiram phase,e tc.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Placebo | Disulfiram 250 | Disulfiram 375 | Disulfiram 500
Number analyzed (Participants) | 27 | 25 | 30 | 25
Weeks | 8.3 (5.4) | 9.0 (4.9) | 6.4 (4.7) | 8.3 (4.8)
Statistical Analysis 1: Comparison: Placebo vs Disulfiram 250 vs Disulfiram 375 vs Disulfiram 500; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.5

ADVERSE EVENTS:
Time Frame: 12 weeks (during disulfiram phase) plus 2 wk washout
Description: although participants were out of the protocol at the end of week 14, because disulfiram could interact with alcohol for up to 2 weeks after stopping use, we continued to monitor participants during this time.
Arm/Group | Placebo | Disulfiram 250 | Disulfiram 375 | Disulfiram 500
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/23 | 1/24 | 0/21
Other Adverse Events (participants affected / at risk) | 8/20 | 12/23 | 10/24 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Disulfiram 250 (N=23) | Disulfiram 375 (N=24) | Disulfiram 500 (N=21)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute COPD exacerbation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal Abcess (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Disulfiram 250 (N=23) | Disulfiram 375 (N=24) | Disulfiram 500 (N=21)
GI Distress (e.g., nausea, vomiting, etc.) (Gastrointestinal disorders) | 2 (2) | 7 (9) | 6 (8) | 6 (6)
Slurred speech (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sweating (General disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Increased Vital Signs (e.g., BP, HR) (Cardiac disorders) | 1 (1) | 4 (5) | 2 (3) | 2 (2)
Metallic or Garlic Taste (General disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Dry mouth/Excessive Thirst (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 3 (3) | 1 (2) | 1 (1)
Lethargy/Sedation (General disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Anxiety/Nervousness (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes